CLINICAL TRIAL: NCT00103155
Title: Radiofrequency Ablation for Low Risk Papillary Thyroid Cancer: A Pilot Study
Brief Title: Radiofrequency Ablation in Treating Patients Who Are Undergoing Surgery for Thyroid Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000410790; UCSF-H28355-23383-01; UCSF-03202
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2005-08

CONDITIONS: Head and Neck Cancer
Keywords: stage I papillary thyroid cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Cancer, Papillary | interventions — Radiofrequency Ablation

INTERVENTIONS:
Procedure: conventional surgery
Procedure: radiofrequency ablation

SUMMARY:
RATIONALE: Radiofrequency ablation uses a high-frequency, electric current to kill tumor cells. Ultrasound-guided radiofrequency ablation may be effective treatment for thyroid cancer.

PURPOSE: This phase I trial is studying the side effects of radiofrequency ablation in treating patients who are undergoing surgery for thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency of complications associated with radiofrequency ablation (RFA) in patients with low-risk papillary thyroid cancer undergoing thyroidectomy.
* Determine the utility of RFA as a treatment option for these patients.

OUTLINE: This is a pilot study.

An electrosurgical probe is placed by ultrasound guidance into the center of the thyroid tumor. Patients undergo radiofrequency ablation directly to the tumor until the target temperature is reached* for 5 minutes. Patients then undergo standard thyroidectomy.

NOTE: *Takes approximately 15-30 minutes to reach target temperature.

After completion of study treatment, patients are followed at day 1, between days 14-21, and then periodically as deemed necessary.

PROJECTED ACCRUAL: A total of 15-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically confirmed papillary thyroid cancer by fine needle aspiration

  * Low-risk disease
  * No poorly differentiated cytology
* Intrathyroidal tumor

  * Located within the anterior two-thirds of the thyroid lobe
  * Tumor not adjacent to the trachea by neck ultrasound
* Tumor ≤ 1.5 cm by neck ultrasound
* Requires thyroidectomy
* No cervical lymphadenopathy
* No multicentric tumors by neck ultrasound
* No evidence of lymph node metastasis

PATIENT CHARACTERISTICS:

Age

* Over 21

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-09

PRIMARY OUTCOMES:
Frequency of radiofrequency ablation-associated complications at 2 weeks

SECONDARY OUTCOMES:
Amount of tumor destruction at 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Electron Kebebew, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States